CLINICAL TRIAL: NCT00063791
Title: An Open-Labeled, Randomized Study to Assess Two Different Strategies of Combining Dexamethasone and VELCADE in Patients With Relapsed Multiple Myeloma Who Have Failed Four or More Lines of Therapy
Brief Title: A Study to Assess Two Different Strategies of Combining Dexamethasone and VELCADE
Status: No longer available | Type: Expanded Access
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Other Study IDs: M34102-052
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2003-07

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
The purpose of this study is to give patients who have had 4 or more prior lines of therapy for multiple myeloma access to VELCADE. The study is for patients who are not eligible for other clinical trials with VELCADE and for who VELCADE would otherwise not be available.

ELIGIBILITY:
Inclusion Criteria:

Major Criteria:

* Plasmacytomas on tissue biopsy
* Bone marrow plasmacytosis (> 30% plasma cells)
* Monoclonal IgG is > 3.5 g/dL or IgA is > 2.0 g/dL; kappa or lambda light chain excretion is > 1 g/day on a 24 hour urine sample.

Minor criteria:

* Bone marrow plasmacytosis (10 to 30%)
* Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria.
* Lytic bone lesions

Other Eligibility Requirements:

* Patient is not eligible for Millennium Study M34101-039.
* Patient has received 4 or more lines of therapy for multiple myeloma and, in the investigator's opinion, currently needs therapy because of relapsed or progressive disease.
* Patient is of legal consenting age, as defined by local regulations.
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Female patients must be either post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control throughout the study.
* Male patients must agree to use an acceptable method of birth control throughout the study.
* Patient has a Karnofsky performance status of greater than or equal to 60%.
* Patient meets pretreatment laboratory criteria at and within 14 to 21 days before Baseline (Day 1 of Cycle 1, before study drug administration).

Exclusion Criteria:

* Patient progressed while receiving VELCADE previously in a clinical trial.
* Patient has been treated in Millennium Study M34101-039.
* Patient received corticosteroids (> 10 mg/day prednisone or equivalent) within 1 week before enrollment in the study.
* Patient received nitrosoureas within 6 weeks or any other chemotherapy within 3 weeks before enrollment in the study.
* Patient received immunotherapy or antibody therapy within 4 weeks before enrollment.
* Patient had major surgery with 4 weeks before enrollment (kyphoplasty isn't considered major surgery).
* Patient has a history of allergic reactions due to compounds containing boron or mannitol.
* Patient has peripheral neuropathy of Grade 2 or greater, as defined by the National Cancer Institute Common Toxicity Criteria (NCI CTC).
* Patient has a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias or electrocardiogram shows evidence of acute ischemia or active conduction system abnormalities.
* Patient has cardiac amyloidosis
* Patient has poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment.
* Patient is known to be infected with human immunodeficiency virus (HIV positive).
* Patient is known to be hepatitis B positive or has active hepatitis C infection.
* Patient has an active systemic infection requiring treatment.
* Female patient is pregnant or breast-feeding. Confirmation that the patient is not pregnant is required. Pregnancy testing is not required for post-menopausal or surgically sterilized patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Michael Meshad, Oncology Center, Mobile, Alabama
  - Henry Ford Health System, Detroit, Michigan
  - Toledo Clinic, Toledo, Ohio